CLINICAL TRIAL: NCT05031676
Title: Efficiency of Opioid-free Anesthesia (OFA) in Maxillofacial Surgery
Brief Title: Opioid Free Anesthesia in Maxillofacial Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université NAZI BONI (Other)
Responsible Party: Principal Investigator, Ismael Guibla, Anaesthesist, Université NAZI BONI
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: INSSA
Record Dates: First submitted 2021-08-07; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Maxillofacial Surgery

STUDY DESIGN:
Intervention Model Description: The patients were randomized during the pre-anesthetic visit in two groups 1 and 2. They were randomized in blocks of four so that, in each block of four patients, there were two patients for the protocol 1 and two patients for the protocol 2.
Who Masked: Participant
Masking Description: Participant does not know the protocol which receive but i
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Intervention consists at induction : direct intravenous lidocaine 1.5 mg/kg; clonidine 2 μg/kg in 250 ml of isotonic saline, started as soon as the venous route is taken and over a period of approximately 15 minutes; magnesium sulfate 50 mg/kg in the same isotonic saline as clonidine.
  Interventions: Other: opioid free anesthesia
- group 2 (No Intervention): In classic induction: fentanyl at a dose of 2 µg/kg. Following induction in all patients consisted of the administration of propofol 2-3 mg/kg in titration, rocuronium 0.6 mg/kg, ketamine 0.5 mg/kg, methylprednisolone 120 mg.

INTERVENTIONS:
Other: opioid free anesthesia — Maintenance of anesthesia was done with halothane. The incision was allowed at 1.2 MAC of halothane. This halogen was administered according to the hemodynamic parameters and the habits of the anesthesia team. Before waking up, all the patients benefited from preventive analgesia with 1 g paracetamol combined with 20 mg nefopam by slow intravenous injection over approximately 15 minutes.
  Arms: group 1

SUMMARY:
Opioid free anesthesia is a promising practice in anesthesia. Studies already carried out have compared OFA to an opioid or "opioid anesthesia" (OA) protocol without the use of antihyperalgesic in the OA protocol. Most of the studies currently available have been carried out in Europe, America and a few in Asia under conditions other than those available in precarious situations.That's why we decide to conduct a study to evaluate the effectiveness of an OFA protocol in maxillofacial surgery in Burkina Faso.

DETAILED DESCRIPTION:
The patients were recruited at the University Hospital of Souro Sanou in Bobo Dioulasso

ELIGIBILITY:
Inclusion Criteria:

* All patients aged between 15 and 65 years, admitted to the central operating room of the hospital for maxillofacial surgery.

Exclusion Criteria:

* Known or suspected coronary artery disease on preoperative consultation;
* Unstable arterial hypertension
* Insulin-dependent diabetes
* Second degree atrioventricular block
* Neuro-vegetative dysautonomia;
* known allergy or intolerance to a drug of the protocols

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Highest numerical pain score | First two hours postoperatively
  The main highest numerical pain score postoperatively

SECONDARY OUTCOMES:
Blood pressure | six minutes after incision
  Changes in blood pressure
Ephedrine | During anesthesia
  Intraoperative consumption of ephedrine
Wake up | Time between the end of surgery and extubation
  wake up time
Nausea-Vomiting | During 24 after surgery
  The proportion of nausea-vomiting after surgery
Highest numerical pain score 24 hours | The first 24 hours postoperatively
  The mean of the highest EN score during the first 24 hours postoperatively
Non-surgical complications | During 24 hours after surgery
  The proportion of non-surgical complications within 24 hours of anesthesia
Heart rate | six minutes after incision
  Changes in heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Guibla, Doctor, Principal Investigator — University Hospital Souro Sanou, Burkina Faso; Charles Ilboudo, Doctor, Study Chair — University Hospital Souro Sanou, Burkina Faso; Bertille Ki, Professor, Study Chair — Univesity of Joseph KI-ZERBO, Health sciences institute; Jean Paul Lechat, Doctor, Study Chair — Hospital of Charleroi (GHdC), Belgium; Cheick Bougouma, Doctor, Study Chair — Univesity of Joseph KI-ZERBO, Health sciences institute; Alain Traore, Professor, Study Director — University of Nazi Boni, Health sciences institute; Flavien Kabore, Professor, Study Director — Univesity of Joseph KI-ZERBO, Health sciences institute
Locations (1):
- Guibla, Bobo-Dioulasso, Houet, Burkina Faso

IPD SHARING:
Plan to Share IPD: No
Use number and date to find participant folder. Participant data are confidential.

REFERENCES:
- [Result] De Kock M. L'anesthésie sans opiacés : anecdote ou nécessité ? Douleur et Analgésie. 2014 sept;27(3):145-148.
- [Result] Beloeil H. Anesthésie sans opiacés. Anesth Réanimation. 2018 may;4(3):215-218.
- [Result] Mulier J. Opioid free general anesthesia: A paradigm shift? Rev Esp Anestesiol Reanim. 2017 Oct;64(8):427-430. doi: 10.1016/j.redar.2017.03.004. Epub 2017 Apr 18. No abstract available. English, Spanish. PMID 28431750
- [Result] Parsa FD, Cheng J, Stephan B, Castel N, Kim L, Murariu D, Parsa AA. Bilateral Breast Reduction Without Opioid Analgesics: A Comparative Study. Aesthet Surg J. 2017 Sep 1;37(8):892-899. doi: 10.1093/asj/sjx038. PMID 28333299
- [Result] Mansour MA, Mahmoud AA, Geddawy M. Nonopioid versus opioid based general anesthesia technique for bariatric surgery: A randomized double-blind study. Saudi J Anaesth. 2013 Oct;7(4):387-91. doi: 10.4103/1658-354X.121045. PMID 24348288
- [Result] Soffin EM, Wetmore DS, Beckman JD, Sheha ED, Vaishnav AS, Albert TJ, Gang CH, Qureshi SA. Opioid-free anesthesia within an enhanced recovery after surgery pathway for minimally invasive lumbar spine surgery: a retrospective matched cohort study. Neurosurg Focus. 2019 Apr 1;46(4):E8. doi: 10.3171/2019.1.FOCUS18645. PMID 30933925
- [Result] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. [Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study]. Rev Bras Anestesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjan.2014.05.006. Epub 2014 Nov 1. Portuguese. PMID 25990496
- [Result] Toleska M, Dimitrovski A. Is Opioid-Free General Anesthesia More Superior for Postoperative Pain Versus Opioid General Anesthesia in Laparoscopic Cholecystectomy? Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2019 Oct 1;40(2):81-87. doi: 10.2478/prilozi-2019-0018. PMID 31605587